CLINICAL TRIAL: NCT00597337
Title: Using a Virtual Learning Environment to Reduce Bullying: Evaluation of the FearNot!v.2.0 Intervention in Primary Schools in England and Germany
Brief Title: Effectiveness of the FearNot!v.2.0 Software in Reducing Bullying Victimisation Among Primary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Warwick (Other)
Collaborators: University of Wuerzburg (Other); University of Hertfordshire (Other); University of Bamberg (Other); European Commission (Other)
Responsible Party: Professor Dieter Wolke, University of Warwick
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WAR-IST-4-027656-STP; IST-4-027656-STP
Record Dates: First submitted 2008-01-09; First posted 2008-01-18 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-10

CONDITIONS: Bullying Victimisation
Keywords: bullying; victimisation; aggressive behavior
MeSH Terms: conditions — Bullying; Aggression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Receiving FearNot
  Interventions: Behavioral: FearNot
- 2 (No Intervention): Control: Treatment as usual (normal curriculum)

INTERVENTIONS:
Behavioral: FearNot — Behavioral: Three sessions of FearNot!v.2.0 software interaction over a three-week period (each session lasting approximately 30 minutes)
  Arms: 1

SUMMARY:
This study will evaluate the effectiveness of a virtual learning treatment in reducing bullying among primary school children in the UK and Germany.

DETAILED DESCRIPTION:
In this study, a virtual learning environment application called FearNot!v.2.0 will be evaluated as a way to improve the quality of life in schools by altering children's attitudes and behavior towards bullying.

Participants will be assigned to either the intervention or the control group. The intention was to assign randomly, however, only a minority of primary schools have the computer facilities to run the software with all pupils participating. Thus, assignment is based on the school computer compatibility with the FearNot!v.2.0 software for intervention versus control group controlling for social variables. Participants in the intervention group will interact with the software during 30-minute sessions once a week for a total of 3 weeks while participants in the control group will follow the normal curriculum.

The FearNot! narrative comprises a number of emergent episodes, which play out like an improvisational drama. During each of these emergent episodes, the characters will act out their roles resulting in a dramatic movie-like display on the computer's monitor. In between each of these episodes, the child can interact with the victim character. He/she can learn how the character feels, and offer them coping strategy advice as to how to behave in the following episode.

Outcomes will be assessed through student questionnaires at baseline, one week, and four weeks after treatment. In addition, classroom teachers will be asked to complete the Teacher Incidence of Bullying Scale at baseline and 4 weeks after the treatment.

ELIGIBILITY:
Inclusion Criteria for schools:

* Mixed
* Not currently involved in intervention studies specific to countering bullying
* Access to computers that are compatible to run FearNot!v.2.0 (for intervention schools)

Inclusion Criteria for participants:

* Age between 8-11
* Passive parental consent

Exclusion Criteria:

* Enrolled in special education schools

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1129 (Actual)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Bullying victimisation - Participant Roles Questionnaire | Measured 1 week post-treatment and at 4 week follow-up

SECONDARY OUTCOMES:
Knowledge about Bullying and Coping Strategies Knowledge Questionnaire | Measured 1-week post-treatment and at 4-week follow-up
Peer nominations of defenders | Measured 1 week post-treatment and at 4 week follow-up
Hymel, Rocke & Bonanno Moral Disengagement Questionnaire | Measured 1 week post-treatment and at 4 week follow-up
Janke and Janke Adjective Word List (adapted) | Measured after each treatment session

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Wolke, PhD, Principal Investigator — University of Warwick
Locations (1):
- University of Warwick, Coventry, United Kingdom

REFERENCES:
- [Derived] Sapouna M, Wolke D, Vannini N, Watson S, Woods S, Schneider W, Enz S, Hall L, Paiva A, Andre E, Dautenhahn K, Aylett R. Virtual learning intervention to reduce bullying victimization in primary school: a controlled trial. J Child Psychol Psychiatry. 2010 Jan;51(1):104-12. doi: 10.1111/j.1469-7610.2009.02137.x. Epub 2009 Aug 24. PMID 19703096